CLINICAL TRIAL: NCT01293669
Title: Phase II Study of Glycemic Control, Safety, Tolerability and Pharmacokinetic Parameters of TC-6987 Monotherapy in Subjects With Type 2 Diabetes Mellitus
Brief Title: Glycemic Control, Safety and Tolerability of TC-6987 Monotherapy in Type 2 Diabetes Mellitus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Targacept Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC-6987-23-CRD-002
Record Dates: First submitted 2011-02-09; First posted 2011-02-10 (Estimated); Last update posted 2013-09-13 (Estimated); Status verified 2012-07

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 Diabetes; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- TC-6987 (Experimental)
  Interventions: Drug: TC-6987
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: TC-6987 — TC-6987-23 (TC-6987 HCl) as experimental treatment: 20 mg loading dose (2 capsules) on Day 1 and 10 mg (1 capsule) on Days 2 to 28 (dose expressed as free base). Each dose will be given once daily.
  Arms: TC-6987
Drug: Placebo — Matching placebo: Mode of administration: p.o. (microcrystalline cellulose in capsule) given once daily.
  Arms: Placebo

SUMMARY:
TC-6987 is a selective nicotinic α-7 receptor ligand (open channel stabilizer) that has demonstrated potent anti-inflammatory/antioxidant properties in animal models. Following the oral administration of a 1mg/kg dose of TC-6987 to diabetic mice (db/db mouse) for 7 weeks, numerous metabolic improvements were observed. Specifically, plasma glucose and triglyceride concentrations declined by approximately 30%; Hb1Ac was reduced by nearly 50%; and TNF-α declined more than 60% relative to control db/db mice Therefore, it appears that TC-6987 could prove beneficial in reducing elevated glucose concentrations in diabetic patients as well as in ameliorating organ damage associated with inflammation, oxidative stress and hyperglycemia.

DETAILED DESCRIPTION:
This is a Phase II, multicenter, randomized, double-blind, parallel group, placebo-controlled study to assess the efficacy, safety, tolerability, and pharmacokinetic parameters of TC-6987 in subjects with type 2 diabetes mellitus (T2DM). The study is organized into three phases: (a) Screening phase consisting of a 1-week Screening (Week -5)and a 4-week Washout (Week -4 to Day 1); (b) 4-week, Double-Blind Treatment (Day 1 to Week 4) during which subjects are randomized to either TC-6987 (20 mg on Day 1 and 10 mg from Day 2 to Week 4) or placebo; and (c) 2-week Follow-Up (Week 6). Unscheduled visits will be allowed between visits from Washout through Follow-up to evaluate a subject's glycemic status or other safety issues, as required. Subjects will fast overnight for a minimum of 10 hrs and refrain from drinking alcohol 24 hrs prior to each visit.

ELIGIBILITY:
Inclusion Criteria:

* Males or postmenopausal/surgically sterile females
* Being treated for T2DM with oral antidiabetic agents (excluding glitazones)
* BMI limit ≤ 38
* Subjects at least 80% compliant on reporting daily SMBG values during washout
* At the end of washout the subject's fasting SMBG is higher than it was at the start of washout and the fasting SMBG ≤ 280.g treated for T2DM with oral antidiabetic agents (excluding glitazones)

Exclusion Criteria:

* Type 1 diabetes mellitus
* Severe complications of T2DM (especially diabetic retinopathy imminently requiring treatment for preserving or restoring vision, diabetic neuropathy with symptomatic orthostatic hypotension, urinary retention, gastric stasis, or pedal ulcers)
* Current treatment with insulin or a glitazone
* Use of moderate to strong cytochrome P450 3A4 (CYP3A4) inhibitors
* FSH level of < 35 IU/L and a LH level < 25 IU/L except for confirmed surgically sterile women with functioning ovaries
* Significant cardiovascular diseases (including arrhythmia) or congestive heart failure, or severe ischemic disease within the last 3 months prior to Screening, or evidence of stroke, myocardial infarction, unstable angina, coronary bypass and/or percutaneous transluminal coronary angioplasty
* History of significant other major or unstable neurological, metabolic, hepatic, renal, hematological, pulmonary, CV, GI, or urological disorder; or diagnosis of major depressive disorder; if stable medical disorder, any medical treatment must be stable for last 2 months prior to Screening
* History of diabetic ketoacidosis
* Patients who have an increased red blood cell (RBC) turn-over or thalassemia or anemia
* Known HIV or history of viral hepatitis type B or C
* Systemic infection with TB
* Current or previous use of oral or injectable corticosteroids 3 months prior to screening.
* Subject has persistent, uncontrolled severe hypertension as indicated by a systolic blood pressure > 180 mmHg or a diastolic blood pressure of > 110 mmHg, with or without treatment
* Subject has had a malignancy in the last 5 years, except for successfully treated basal or squamous cell carcinoma of the skin or of the cervix
* Subject is receiving chemotherapy
* Tobacco user within 4 months prior to Screening
* Smoking cessation therapy within 4 months prior to Screening and/or planned during the study
* Use of prohibited concomitant medications including psychoactive agents
* History within 6 months prior to Screening of alcohol abuse or illicit drug abuse
* Was administered study medication in another clinical trial in the past 3 months prior to Screening

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 440 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Changes in fasting plasma glucose (FPG) | Day 1 and Week 4
  The primary efficacy endpoint will be FPG values obtained at Week 4 compared to Day 1 (baseline). This change from baseline will be analyzed using MMRM techniques with an alpha of 0.10 (one-sided), to examine differences between the TC-6987 and placebo treatment cohorts. This change from baseline will be analyzed using the primary efficacy endpoints for the mITT analysis set. The efficacy analyses based on the Per Protocol (PP) analysis set will be considered secondary.

SECONDARY OUTCOMES:
Change in FPG from Day 1 (Baseline) at each time point | Day 1, Week 1 and Week 4
  Change in FPG from Day 1 (Baseline) compared to weeks 1 and 4
Change in FPG and insulin from Day 1 (Baseline) at each time point | Day 1, Week 1 and Week 4
  Change in FPG and insulin from Day 1 (Baseline) compared to weeks 1 and 4
Change in AUC FPG from Day 1 (Baseline) and at Week 4 | Day 1 and Week 4
  Change in AUC FPG from Day 1 (Baseline) compared to weeks 1 and 4
Change in AUC insulin from Day 1 (Baseline) at Week 4 | Day 1 and Week 4
  Change in AUC insulin from Day 1 (Baseline) compared to week 4

CONTACTS AND LOCATIONS:
Overall Officials: Aaron Vinik, MD, Principal Investigator — Strelitz Diabetes Center, Eastern Virginia Medical School
Locations (18):
- United States (18):
  - Clopton Clinic, Jonesboro, Arkansas
  - NCA Medical Center, Mountain Home, Arkansas
  - Associated Pharmaceutical Research Center, Buena Park, California
  - Cedar Crosse Research Center, Chicago, Illinois
  - Medex Healthcare Research, Inc, St Louis, Missouri
  - Om Medical, Henderson, Nevada
  - MEDEX Healthcare Research, Inc, New York, New York
  - PMG Research of WS, Winston-Salem, North Carolina
  - Rapid Medical Research, Inc., Cleveland, Ohio
  - Providence Health Partners - Center for Research, Dayton, Ohio
  - Omega Medical Research, Warwick, Rhode Island
  - Ellipsis Research, Columbia, South Carolina
  - PMG Research of Charleston, Mt. Pleasant, South Carolina
  - New Phase Research and Development, Knoxville, Tennessee
  - Mercury Clinical Research, Houston, Texas
  - Quality Research, Inc., San Antonio, Texas
  - Highland Clinical Research, Salt Lake City, Utah
  - Strelitz Diabetes Center, Eastern Virginia Medical School, Norfolk, Virginia